CLINICAL TRIAL: NCT02509182
Title: The Effect of Decreasing the Inspired Oxygen Concentration on Post-Operative Oxygenation After Primary Lobectomy: A Randomized Controlled Trial
Brief Title: The Effect of Decreasing the Inspired Oxygen Concentration on Post-Operative Oxygenation After Primary Lobectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never officially began
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1507016157
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Hyperoxia
Keywords: Hyperoxia; One-Lung Ventilation; Thoracic Surgery; Anesthesiology
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100% FiO2 (Active Comparator): 100% oxygen administered during pulmonary lobectomy surgery.
  Interventions: Drug: 100% oxygen
- 60% FiO2 (Experimental): 60% oxygen administered during pulmonary lobectomy surgery.
  Interventions: Drug: 60% oxygen

INTERVENTIONS:
Drug: 60% oxygen — An inspired oxygen concentration of 60% will be administered during pulmonary lobectomy surgery.
  Other Names: FiO2 60%
  Arms: 60% FiO2
Drug: 100% oxygen — An inspired oxygen concentration of 100% will be administered during pulmonary lobectomy surgery.
  Other Names: FiO2 100%
  Arms: 100% FiO2

SUMMARY:
The purpose of this study is to test the hypothesis that decreasing the inspired oxygen concentration during thoracic surgery requiring one lung ventilation will improve post-operative oxygenation.

DETAILED DESCRIPTION:
One lung ventilation is frequently required during thoracic surgery and results in decreased lung function post-operatively. Supra-physiologic oxygen levels during surgery may contribute to this decrease in lung function by worsening lung injury intra-operatively.

This study will include patients undergoing surgery to remove a lung lobe requiring one lung ventilation.

The patients will be divided into two groups with the experimental group receiving a 60% oxygen in air mixture and the control group receiving 100% oxygen.

The two groups will be compared by using a measure of lung function (the ratio of the partial pressure of oxygen in arterial blood to the inspired oxygen concentration) and blood levels of a protein correlated with lung injury (receptor of advanced glycation end products RAGE).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age and older, male or female.
2. American Society of Anesthesiology (ASA) physical status I, II, III or IV
3. Subjects who are scheduled for elective primary pulmonary lobectomy.
4. Subjects who have an arterial line placed as part of routine anesthetic management
5. Subjects who can understand and communicate in English.

Exclusion Criteria:

1. Subjects with a history of difficult intubation
2. Subjects with a high risk of aspiration during induction of anesthesia
3. Subjects with morbid obesity (BMI greater than or equal to 40)
4. Subjects with unable to provide consent
5. Subjects who are minors
6. Subjects who are not English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
PaO2 to FiO2 ratio | Post-operative day 1
  The ratio of the partial pressure of oxygen in arterial blood (PaO2) to the inspired oxygen concentration (FiO2). An arterial blood sample will be drawn from an arterial line on post-operative day 1 and the FiO2 at the time of blood draw will be documented to calculate the ratio.

SECONDARY OUTCOMES:
Mortality | 30 days
  Mortality will be determined by accessing the medical record.
Mortality | 1 year
  Mortality will be determined by accessing the medical record.
Hypoxemia less than 90% | Intra-operative
  This will be recorded from the intraoperative data acquired during surgery.
Blood level of receptor of advanced glycation end-products (RAGE) protein | Post-operative day 1
  The receptor of advanced glycation end-products (RAGE) protein levels correlates with alveolar epithelial lung cell injury and will be measured in a blood sample collected on post-operative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Popescu, MD, Principal Investigator — Yale University; Nathan Clendenen, MD,MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States